CLINICAL TRIAL: NCT04017104
Title: A Sub-study of 18F-DCFPyL Positron Emission Tomography / Computed Tomography (PET/CT) for Assessment of Recurrent Prostate Cancer Evaluation of the Safety and Sensitivity of 68Ga-DOTATOC PET/CT for Imaging NET Patients
Brief Title: Dynamic Whole Body Positron Emission Tomography/Computed Tomography Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H19-00623
Record Dates: First submitted 2019-05-27; First posted 2019-07-12 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Neuroendocrine Tumors; Prostate Cancer; Prostatic Neoplasms; Carcinoid Tumor; Paraganglioma; Neuroblastoma
MeSH Terms: conditions — Neuroendocrine Tumors; Prostatic Neoplasms; Carcinoid Tumor; Paraganglioma; Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 18F-FDG PET/CT Diagnostic Imaging: Participants that have been chosen and consented to participate in the optional DWB PET/CT scan sub-study will undergo an extra 18F-FDG PET/CT procedure.
  18FFDG is considered standard care and has been approved by Health Canada.
  Interventions: Diagnostic Test: 18F-FDG PET/CT
- 68Ga-DOTATOC PET/CT Diagnostic Imaging: Participants that have been chosen and consented to participate in the optional DWB PET/CT scan sub-study will undergo an extra 68Ga-DOTATOC PET/CT procedure.
  The 68Ga-DOTATOC radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada.
  Interventions: Diagnostic Test: 68Ga-DOTATOC PET/CT
- 18F-DCFPyL PET/CT Diagnostic Imaging: Participants that have been chosen and consented to participate in the optional DWB PET/CT scan sub-study will undergo an extra 18F-DCFPyL PET/CT procedure.
  The 18F-DCFPyL radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada.
  Interventions: Diagnostic Test: 18F-DCFPyL PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT — For 18F-FDG as fasting period of 6 hours is required before the scan. Each study subject will have an intravenous catheter inserted. The subject will receive a bolus intravenous dose of the radiotracer from an approved study supplier site.The participant will rest in a comfortable chair for 20 minutes. The participant will then be taken to a designated washroom and asked to void prior to being scanned in order to clear excreted radiotracer activity from the urinary tract. The participant will then be taken to the PET/CT scanner.
  Subjects are positioned supine, arms down, and centered on the scanner bed and the PET/CT images will be acquired.
  Groups: 18F-FDG PET/CT Diagnostic Imaging
Diagnostic Test: 68Ga-DOTATOC PET/CT — Participants will not be encouraged to drink additional water due to the requirement to stay on the scanner for up to 90 minutes. There are no dietary restrictions. Each study subject will have an intravenous catheter inserted. The participants will then be taken to a designated washroom and asked to void, and will then be taken to the PET/CT scanner. A CT topogram will be acquired followed by very low dose whole body CT for attenuation correction and localization of PET emission data. The participant will receive a bolus intravenous dose of the radiotracer 68Ga-DOTATOC from an approved study supplier site. Simultaneously a 6 minute dynamic acquisition of the heart will be started, then followed by several whole body static acquisitions. After the DWB scan, participants may go to the washroom again and their vital signs will be recorded. After this, a new PET/CT acquisition, as specified in the 68Ga-DOTATOC PET/CT protocol, will immediately follow.
  Groups: 68Ga-DOTATOC PET/CT Diagnostic Imaging
Diagnostic Test: 18F-DCFPyL PET/CT — Participants will not be encouraged to drink additional water due to the requirement to stay on the scanner for 90 minutes of the DWB acquisition. They will be unable to use the washroom during this time. As with the main study, participants will be instructed to fast for 4 hours prior to their appointment. Each study subject will have an intravenous catheter inserted. The participants will then be taken to a designated washroom and asked to void, and will then be taken to the PET/CT scanner. The participant will receive a bolus intravenous dose of 18F-DCFPyL from an approved supplier. This will then be followed by several whole body static acquisitions for a total scan time that will not be longer than 90 minutes. After the scan is finished, the participant will be allowed to rest in a comfortable chair or bed for 30 minutes. The participants will return to the scanner room and undergo the planned PET/CT imaging described in the main study.
  Groups: 18F-DCFPyL PET/CT Diagnostic Imaging

SUMMARY:
Quantitative parameters obtained with dynamic whole body imaging using positron emission tomography (PET) can provide additional and complementary information to standard PET. Dynamic imaging allows for better understanding of the behavior of the radio-pharmaceutical because it can be followed over time. Thought to be difficult to perform with currently available clinical equipment that can affect the clinical workflow, it has recently shown to be feasible. We want to test the feasibility of this imaging technique and evaluate its utility in identifying lesions with three different radio-pharmaceuticals as compared to standard static PET.

This study will also determine the clinical impact of DWB PET on participant management by comparing the overall qualitative assessment performed by nuclear medicine physicians between the standard PET images and the DWB ones.

DETAILED DESCRIPTION:
This is a prospective single cohort study to evaluate the feasibility of dynamic whole body PET/CT in identifying and quantifying lesions where standard static PET has been negative or equivocal.

18F-FDG PET/CT - Participants that have been chosen and consented to participate in the optional DWB PET/CT scan sub-study will undergo an extra 18F-FDG PET/CT procedure. 18F-FDG is considered standard care and has been approved by Health Canada. A fasting period of 6 hours is required before the scan. Diabetic participants should withhold short acting insulin during the fasting interval, and discuss with their physician whether to reduce long acting insulin the morning of the examination. Participants will also be instructed to drink 3 to 4 glasses of water within two hours prior to their scan appointment in order to promote hydration and facilitate urinary clearance of background radiopharmaceutical.

Prior to the 18F-FDG PET/CT procedure, participants will be instructed to take their usual medications as prescribed by their physician.

After providing informed written consent subjects will complete a medical history questionnaire.

The PET dynamic scan will start 30 minutes after the 18F-FDG injection. This will be followed by several whole body static acquisitions for a total scan time that will not be longer than 32 minutes.

After the DWB scan is finished, participants will be given the option to go to the washroom again. After this, a new PET/CT acquisition, as specified in the 18F-FDG PET/CT scan protocol, will immediately follow. Upon completion of the second PET scan, participants will be free to leave the department and will be encouraged to drink 3 - 4 extra glasses of water by the end of the day to promote further clearance of the remaining tracer in the urinary tract.

68Ga-DOTATOC PET/CT - Participants that have been chosen and consented to participate in the optional DWB PET/CT scan sub-study will undergo an extra 68Ga-DOTATOC PET/CT procedure. The 68Ga-DOTATOC radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada. Prior to the 68Ga-DOTATOC PET/CT procedure, participants will be instructed to take their usual medications as prescribed by their physician. After providing informed written consent subjects will complete a medical history questionnaire. Participants will not be encouraged to drink additional water due to the requirement to stay on the scanner for up to 90 minutes (60 min DWB followed by standard PET acquisitions). There are no dietary restrictions.

After the DWB scan is finished, participants will be given the option to go to the washroom again and their vital signs will be recorded one more time. For this sub-study the vital signs will not be collected after the radiotracer injection to accommodate for the DWB protocol. After this, a new PET/CT acquisition, as specified in the 68Ga-DOTATOC PET/CT protocol, will immediately follow. Upon completion of the second PET scan, participants will be free to leave the department and will be encouraged to drink 3 - 4 extra glasses of water by the end of the day to promote further clearance of the remaining tracer in the urinary tract.

18F-DCFPyL PET/CT - Participants that have been chosen and consented to participate in the optional DWB PET/CT scan sub-study will undergo an extra 18F-DCFPyL PET/CT procedure. The 18F-DCFPyL radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada.After providing informed written consent subjects will complete a medical history questionnaire. Prior to the 18F-DCFPyL PET/CT procedure, participants will be instructed to take their usual medications as prescribed by their physician. Participants will not be encouraged to drink additional water due to the requirement to stay on the scanner for 90 minutes of the DWB acquisition. They will be unable to use the washroom during this time. As with the main study, participants will be instructed to fast for 4 hours prior to their appointment. The participant will receive a bolus intravenous dose of 18F-DCFPyL from an approved supplier, at a dose of approximately 296 MBq followed by a 5 to 20 mL normal saline flush and simultaneously a 6 minute dynamic acquisition of the heart will be started. This will then be followed by several whole body static acquisitions for a total scan time that will not be longer than 90 minutes.After the DWB scan is finished, the participant will be allowed to rest in a comfortable chair or bed for 30 minutes. During this time the vital signs will be recorded again. For this sub-study the vital signs will be measured before the radiotracer injection and again after the DWB PET scan to accommodate the DWB protocol. The participants will then be taken to a designated washroom and asked to void prior to the standard PET scan to clear excreted 18F-DCFPyL activity from the urinary tract.The participants will return to the scanner room and undergo the planned PET/CT imaging described in the main study.

Participant adverse event monitoring will be completed as part of regular standard of care (18F-FDG) or according to the main study protocols.

Follow-up Assessments - Follow-up information will be collected from the patient's medical records for up to 5 years following the PET/CT scan to obtain confirmatory information (from pathology and additional imaging showing progression or regression under treatment) about the status of known lesions.

The study is expected to take approximately 4 years for accrual.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Meet the inclusion criteria for the appropriate main study (68Ga-DOTATOC PET/CT or 18F-DCFPyL PET/CT) or standard of care imaging.
* Able to not use the washroom for the duration of the dynamic imaging scanning.
* World health organization performance status 0-2
* Able to provide written informed consent/assent (or consent by guardian for subjects <19 years)
* Patients must be able to tolerate the physical/logistical requirements of completing a PET scan including lying flat for up to 30 minutes and tolerating intravenous cannulation for injection.

Exclusion Criteria:

* Pregnancy
* Unable to provide written consent
* Patients who are medically unstable ex: acute cardiac or respiratory distress, hypotensive
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT bore (diameter 70cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to evaluate the diagnostic utility of DWB PET/CT in identifying and quantifying lesions where standard PET imaging (i.e. static) have been negative or equivocal.
  Concordance with histology, imaging or follow-up, using the data collected in the main studies, will also be assessed. This study will also determine the clinical impact of DWB PET on participant management by comparing the overall qualitative assessment performed by nuclear medicine physicians between the standard PET images and the DWB ones.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of dynamic whole body PET/CT imaging with participants: survey | 24 hours
  Feasibility will be measured using a survey that rates participant comfort on a scale from 1 (very uncomfortable) to 5 (very comfortable).

SECONDARY OUTCOMES:
Feasibility of dynamic whole body PET/CT imaging with technologists | 24 hours
  Technologists will record whether there were any challenges with performing the scan. This will be recorded on a YES/NO assessment form.
Feasibility of dynamic whole body PET/CT imaging with clinical value | 2 weeks
  Image assessment will be performed by comparing the number of the 5 most active lesions identified in images that integrate the dynamic imaging portion with the number of the 5 most active lesions found in the standard PET/CT scan. Values will include the number of lesions, and quantitative parameters including lesion size and uptakes values.
Confirm information about status of known lesions - progression or regression of lesions | 5 years
  Follow up information on progression or regression of lesions under treatment, will be collected from the patient's medical records following the PET/CT scan. Lesion size on imaging in millimeters will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada